CLINICAL TRIAL: NCT03827330
Title: Retrospective Chart Review of Candida Fungemia
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999919037; 19-I-N037
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Candida Fungemia
Keywords: Candida Parapsilosis; Candida Auris; Candida Lusitaniae; Candida Glabrata; Candida Albicans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients: Patients who had Candida species growth from blood cultures drawn at the National Institutes of Health

SUMMARY:
Background:

Candida can cause infections. The most common kind of Candida at clinics is C albicans. But other kinds have increased at clinics too. Researchers want to review the records of people who were in previous NIH studies who had Candida. They want to find out what risk factors are associaated with this infection.

Objective:

To study the factors that are associated with Candida fungemia to develop. The factors are clinical features, diagnoses, and previous antifungal therapy.

Eligibility:

People who were in prior NIH studies and had Candida

Design:

Researchers will review the records of 62 NIH participants. The records are from 2004 to 2017. They will look at data such as blood test results, diagnosis, and treatments.

Researchers will only reach out to participants if they get approval from a review board.

This research will probably not reveal data that would be important to participants health. But if it does, researchers will try to contact those participants.

Data will be stored in secure computers. They will be stored with a code that only the study team can link to a participant.

DETAILED DESCRIPTION:
This protocol is a chart review of patients who had Candida species grown from blood cultures drawn at the National Institutes of Health. The study will involve only review of patient records and will not require new specimens or participant contact. The patients whose records will be reviewed in this protocol are/were enrolled on a number of different protocols related to their underlying disease(s). Principal investigators of each protocol have been contacted to request permission to conduct this study, and to verify that none of the original protocols or informed consent documents precludes such a review of clinical data.

ELIGIBILITY:
* The study will involve only review of patient records and will not require new specimens or participant contact. The patients whose records will be reviewed in this protocol are/were enrolled on a number of different protocols related to their underlying disease(s).

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who had Candida species grown from blood cultures drawn at the National Institutes of Health from 2004 until 2017.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

PRIMARY OUTCOMES:
The objective of this protocol is to characterize the clinical features, underlying diagnoses, previous antimicrobial therapy, and previous antifungal therapy associated with the development of Candida fungemia, as well as the enrichment of n... | Duration of study
  The objective of this protocol is to characterize the clinical features, underlying diagnoses, previous antimicrobial therapy, and previous antifungal therapy associated with the development of Candida fungemia, as well as the enrichment of non-albicans species of Candida.

CONTACTS AND LOCATIONS:
Overall Officials: Michail S Lionakis, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States